CLINICAL TRIAL: NCT01533662
Title: Phase 2 Study Evaluating the Prophylactic Phenylephrine Infusion for Preventing Hypotension During Spinal Anesthesia for Lower Limb Orthopedic Surgery in the Elderly Patients
Brief Title: Prophylactic Phenylephrine Infusion for Preventing Hypotension During Spinal Anesthesia
Acronym: PPSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0900103
Record Dates: First submitted 2011-06-30; First posted 2012-02-15 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Orthopedic Surgery of Lower Limb
Keywords: phenylephrine; hypotension; spinal anesthesia; lower limb orthopedic surgery
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- phenylephrine (Experimental): patients more than 60 years receiving 100micrograms of phenylephrine infusion (2 groups 60-75 years and more than 75 years)
  Interventions: Drug: phenylephrine infusion
- placebo (Placebo Comparator): patients more than 60 years receiving saline infusion (2 groups 60-75 years and more than 75)
  Interventions: Drug: patients receiving saline infusion

INTERVENTIONS:
Drug: phenylephrine infusion — patients from 60 to 75 years receiving 100micrograms of phenylephrine infusion
  Arms: phenylephrine
Drug: patients receiving saline infusion — patients more than 60 years receiving 100micrograms of saline infusion
  Arms: placebo

SUMMARY:
Lower limb orthopedic surgery is commonly realized under spinal anesthesia. This loco-regional anesthesia induces a peripheral vascular resistance decrease by vasodilatation resulting in hypotension. A severe and prolonged hypotension can compromise regional perfusion and worse outcome especially in very elderly patients. Moreover the venous vasodilatation observed after spinal anesthesia decreases cardiac preload resulting in a cardiac output decrease. Several authors had identified the prevention of hypotension as a key role during spinal anesthesia although none prophylactic treatment has been identified. Spinal anesthesia single injection (SA) with low dose of local anesthetic or continuous spinal anesthesia with very low dose bolus injections cause fewer episodes of hypotension. Despite these techniques, hypotension can occur. Phenylephrine is an alpha adrenergic agonist and cause vasoconstriction preventing hypotension. Prophylactic phenylephrine infusion for preventing hypotension has been demonstrated during spinal anesthesia for cesarean delivery. The investigators want to assess for the first time the prophylactic phenylephrine infusion for preventing hypotension in elderly patients undergoing orthopedic lower limb surgery under spinal anesthesia single injection.

DETAILED DESCRIPTION:
The aim of this study is to assess the prophylactic phenylephrine infusion for preventing hypotension in elderly patients.

This prospective double blinded randomized control trial will include elderly patients over 60 years undergoing orthopedic lower limb surgery under spinal anesthesia single injection (10 mg of Bupivacaine 0,5% with 5 µg of Sufentanyl). We define 4 groups: (1) Patients from 60 to 75 years receiving 100 µg/min of phenylephrine infusion; (2) patients from 60 to 75 years receiving saline infusion; (3) patients over 75 years receiving 100 µg/min of phenylephrine infusion; (4) patients over 75 years receiving saline infusion. Standard monitoring is applied including noninvasive arterial blood pressure, electrocardiography and pulse oximetry. The vasopressor solution and the saline solution will be prepared in identical 50 mL syringes by an investigator not involved in patient care. The investigator administering the solution and the patient are blinded to the content of the syringe. The velocity of infusion will be the same between groups (1ml/min) and the infusion will start once the spinal anesthesia realized. Arterial blood pressure measurements are realized each 1 minute for the first 20 minutes and then each 5 minutes until the end of surgery. After each measurement of MAP, the infusion is stopped if the MAP is more than baseline, and it is continued or restarted if the MAP is less than or equal to baseline. Anyway the infusion is stopped at the end of motor block. Hypotension is defined as a 20% decrease of mean arterial pressure (MAP). Severe hypotension is defined as a 30% decrease of MAP. Hypertension is defined as MAP > 120% of baseline. Each time there is a MAP measurement showing hypotension while patients are under infusion, a 1 mL IV bolus of phenylephrine 100µg/ml is injected by the anesthesiologist involved in patient care. The total volume of study solution given by infusion and the total volume of phenylephrine given by bolus are recorded.

We want to demonstrate fewer episodes of hypotension and fewer post operatory cardiovascular and neurologic events in the groups receiving prophylactic phenylephrine infusion.

ELIGIBILITY:
Inclusion Criteria:

* over 60 years old
* informed consent
* lower limb orthopaedic surgery
* spinal anesthesia

Exclusion Criteria:

* dementia
* anemia less than 10grams per deciliter
* hypertension
* hemostasis disorders
* infection at the puncture
* allergy to local anesthetic,
* patient under anticoagulant.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
number of hypotension episodes | 48h after infusion
  at the end of solution infusion

SECONDARY OUTCOMES:
number of episodes of severe hypotension | 48h after infusion
  at the end of solution infusion
cardiovascular events | 48h after infusion
  at the end of the solution infusion
neurologic events | 48h after infusion
  at the end of solution infusion

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Minville, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, Toulouse, France